CLINICAL TRIAL: NCT02213640
Title: Potentiation of the Effects of Prismatic Adaptation by Transcranial Direct Current Stimulation (tDCS) : Evaluation of Functional Interest in Negligence Rehabilitation
Acronym: PRIStiM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-803
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Neurologic Neglect Syndrome
Keywords: Neurologic neglect syndrome; post stroke; transcranial direct current stimulation (tDCS); prismatic adaptation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A Anodal tDCS and prismatic adaptation (Experimental): anodal tDCS over the primary motor cortex : stimulation intensity of 1mA during 20 minutes (5 consecutive sessions during one week).
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Arm B: control (Placebo Comparator): Prismatic adaptation with placebo stimulation
  Interventions: Device: Control: placebo stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Anodal tDCS over the primary motor cortex. Stimulation intensity of 1mA during 20 minutes (5 consecutive sessions during one week).
  Arms: Arm A Anodal tDCS and prismatic adaptation
Device: Control: placebo stimulation — electrode of sham tDCS over the primary motor cortex during 20 minutes (5 consecutive sessions during one week).
  Arms: Arm B: control

SUMMARY:
Following stroke, over 50% of patients keep severe neurological deficiency whose unilateral neglect, mostly following a right hemispheric lesion. The prismatic adaptation involves to pointing movements toward visual targets wearing prismatic glasses. These prismatic glasses induce a shift to the right visual field for improving symptoms in short term.

Transcranial direct stimulation (tDCS) has been evaluated for different types of deficiency resulting from stroke with encouraging results. The hypothesis of the study is to evaluate the usefulness of brain stimulation as an adjunctive intervention to optimize and increase the rehabilitation of unilateral neglect to long-term.

Thus, the main objective is to evaluate the effectiveness of standard treatment with prismatic adaptation with anodal tDCS or sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* All subjects must be between the ages of 18-80
* Patient with unilateral negligence consecutive to a right hemispheric stroke
* Hospitalized in the Department of Physical Medicine and Rehabilitation (day or week) or external monitoring
* Ischemic or hemorrhagic stroke with right hemispheric topography - evidenced by a radiological report
* Diagnosis of negligence evidenced by Behavioural Inattention Test (BIT) : score ≤ 129
* Stroke >1 month prior to study enrollment

Exclusion Criteria:

* Degenerative neurological complaint
* Uncontrolled epilepsy
* Temporo-spatial disorientation
* Language disorders or psychiatric disorders preventing understanding instructions
* History of prior stroke, multiple stroke
* Medical condition not stabilized
* Pregnancy
* Implanted material (pacemaker, defibrillator, cochlear implant, surgical clips, metal object)
* Intra-cranial material
* Unweaned alcoholism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12-26 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Behavioural Inattention Test (BIT) | Change in BIT score between the baseline sessions average and score measured at week 11
  assessed at two baseline sessions before intervention (inclusion and week 3), and after the therapeutic intervention week (week 5), 2 weeks (week 7), 6 weeks (week 11) and 15 weeks (week 20) following the inclusion.

SECONDARY OUTCOMES:
Negligence Battery Test (BTN) | before intervention (week 1 and week 3), and then again following the intervention (week 5), 2 weeks (week 7), 6 weeks (week 11) and 15 weeks (week 20)
  Change in BTN scores between baseline measures before the therapeutic intervention week and scores obtained during each follow-up sessions
Functional independence scale (MIF) | before intervention (week 1 and week 3), and then again following the intervention (week 5), 2 weeks (week 7), 6 weeks (week 11) and 15 weeks (week 20)
  Change in MIF scores between baseline measures before the therapeutic intervention week and scores obtained during each follow-up sessions
Catherine Bergego scale (ECB) | baseline session before intervention (week 1 and week 3), and then again following the intervention (week 5), 2 weeks (week 7), 6 weeks (week 11) and 15 weeks (week 20)
  Change in ECB scores between baseline measures before the therapeutic intervention week and scores obtained during each follow-up sessions
Jamar | baseline session before intervention (week 1 and week 3), and then again following the intervention (week 5), 2 weeks (week 7), 6 weeks (week 11) and 15 weeks (week 20)
  Change in Jamar scores between baseline measures before the therapeutic intervention week and scores obtained during each follow-up sessions

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JACQUIN-COURTOIS, MD-PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital henri Gabriel (Hospices Civils de Lyon), Saint-Genis-Laval, France

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411